CLINICAL TRIAL: NCT01046747
Title: Pre-drilling Pilot Holes for Self-drilling Schanz Pins: Does it Reduce the Incidence of Pin Tract Infection and Pin Loosening?
Brief Title: Pre-drilling or Self Drilling External Fixation Pins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: John R Fowler, M.D., Temple University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB - 12415 Pin Study
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-08

CONDITIONS: Fracture; Dislocation
Keywords: external fixation; pin tract infection; self drilling
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-drill (Active Comparator): These pins will be pre-drilled
  Interventions: Procedure: Placement of external fixation pins
- No pre-drill (Active Comparator): these pins will not be pre-drilled, but will rely on the self drilling function of the pin for insertion
  Interventions: Procedure: Placement of external fixation pins

INTERVENTIONS:
Procedure: Placement of external fixation pins — The fractures will be treated according to standard of care. If the external fixation is to be used as a staging procedure, then this will be removed and an internal fixation procedure will be performed. The pin sites will be checked daily according to standard of care. All individuals involved in the examination of the pin sites will receive a standardized training in the grading of pin tract infection and loosening. Each pin site will be graded individually by three persons to evaluate internal accuracy of our grading. Pin tract infections will be first graded as yes or no, and then graded according to the Modified Joglekar Classification (Grade 0-4, Grade 0: no erythema, no drainage; Grade 1: erythema, no drainage OR no erythema with serous drainage; Grade 2: erythema, serous drainage; Grade 3: erythema, purulent drainage; Grade 4: gross pin loosening). Pin loosening will be evaluated at the time of pin removal and graded as either yes or no.

SUMMARY:
Hypothesis

There is no difference in the incidence of pin tract infection and pin loosening in case of lower extremity external fixators when self-drilling schanz pins are used with or without pre-drilling.

Primary Objective

The primary objective is to determine whether pre-drilling holes for external fixation pin insertion is superior to not pre-drilling holes for external fixation pin insertion in regards to the incidence of pin tract infection and pin loosening.

Secondary Objective

If any difference is found between the two techniques then, we will quantify and qualify those differences. The incidence of pin site infection and pin loosening in general will be determined and will also be stratified for site and size of pin. An attempt to identify risk factors for pin site infection will be made by observing the effect of secondary prognostic factors like mode of injury, diabetes, smoking, compartment syndrome, peripheral vascular disease, neurovascular injury. Interobserver reliability of the grading system for pin infection will also be determined.

DETAILED DESCRIPTION:
Background

The application of external fixation is a commonly performed emergency procedure in orthopaedics for temporary stabilization as well as definitive treatment of fractures. External fixation requires that metal pins be placed into the bone on either side of the fracture. The pins are then connected to an external frame, thus stabilizing the fracture. There is debate over the optimal technique for the insertion of these pins in regards to the need to pre-drill a pilot hole prior to pin insertion.

The technology behind external fixation has evolved greatly over the past thirty years. The original external fixation pins, "Shanz pins," were essentially metal rods with threads and a trocar point. A pilot hole was needed because these pins did not have the capability to create their own hole or path in the bone. Recent advances have lead to the creation of self-drilling/self-tapping pins, which have decreased the number of steps necessary to place the pins and thereby decreased operative time. The external fixators are usually placed as a temporary measure to allow for improvement of soft tissue condition before definitive open reduction and internal fixation. Since many external fixation devices are placed in patients who are critically ill, decreasing operative time is very important.

While saving operative time is essential it is also important that the device serves its purpose without leading to complications in the short term. The major complications related to external fixation are pin site infection and pin loosening. The literature is clear that high temperatures created during pin insertion leads to bone necrosis surrounding the pin, increased infection, and increased rates of loosening. It is unclear if the new generation self-drilling pins create the same amount of necrosis as the older generation of pins. Lab studies have shown increased temperatures with direct drilling with these pins as compared to pin insertion after drilling pilot holes with dedicated drill bits. It is unclear if this increased temperature results in increased rate of loosening or pin site infection in clinical practice.

A thorough literature search has revealed no randomized controlled studies to support the use of these pins without drilling pilot holes before insertion. The current standard of care is undefined and left to surgeon preference. Our study aims to provide guidelines for schanz pin insertion for external fixator application, which may help to reduce the number of pin tract infections suffered by patients and improve outcomes.

Study Design and Treatment Plan

This will be a prospective, randomized, within-subject, single-blind trial to be conducted at Temple University Hospital. Patients who are determined to require an external fixation procedure of the lower extremities due to fracture or dislocation will be considered for enrollment according to the above inclusion criteria. Standard of care for treatment of their fractures will be provided. Once patients have provided informed consent for enrollment in the study, their pins will be randomized in a paired design according to a computer generated randomization schedule. There will be two types of pins, pre-drilled and non pre-drilled. A standard external fixation device requires two pins on each side of the fracture. Each pair of pins will have one each of pre-drilled and not pre-drilled pins, according to the randomization schedule. Therefore, each patient will have two pre-drilled pins and two pins inserted without pre-drilling. Some surgeons may prefer three pins on each side of the fracture/dislocation that is to be immobilized. We will have a randomization protocol for these situations as well.

The computer generated randomization algorithm will be placed in a secure location in sealed opaque envelopes. The operating surgeon will open the envelope prior to pin insertion and follow the randomization schedule as prescribed in the envelope.

A standard technique will be followed. IV antibiotics will be administered within 60 minutes of the starting skin incision. Pin insertion will be done by standard techniques. This involves a 1 cm incision, and blunt dissection. 4.0 mm (calcaneal or metatarsal), 5.0 mm (tibia) or 6.0 mm (femur) pins will be inserted by one of two techniques: (1) self drilling pins are inserted with a power drill directly into the bone; (2) a standard twist drill bit is utilized with a power drill to create a pilot hole, followed by insertion of the self-drilling pin by power drill.

Soft tissue relaxation incisions are made according to standard technique after external fixation assembly, as needed. The pin care protocol will consist of daily pin site cleaning using dilute hydrogen peroxide and dry dressings. Patients with suspected pin site infection will be treated with Keflex 500mg po q 6hr. Patients with an allergy to Keflex will receive Clindamycin 300mg po q 6hr.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-89
2. Fluency in spoken/ written English/ Spanish (consent form in Spanish will be needed)
3. Lower extremity fracture/ dislocation treated with an external fixator

Exclusion Criteria:

1. Prisoners
2. Patients unable to give informed consent
3. Patients who require that pins be placed without skin coverage at the pin site
4. Patients receiving Ilizarov or other circular external fixators with transfixing wires.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
pin tract infection | until pins are removed

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Abouzgia MB, Symington JM. Effect of drill speed on bone temperature. Int J Oral Maxillofac Surg. 1996 Oct;25(5):394-9. doi: 10.1016/s0901-5027(06)80040-8. PMID 8961026
- [Background] Antoci V, Ono CM, Antoci V Jr, Raney EM. Pin-tract infection during limb lengthening using external fixation. Am J Orthop (Belle Mead NJ). 2008 Sep;37(9):E150-4. PMID 18982187
- [Background] Bachus KN, Rondina MT, Hutchinson DT. The effects of drilling force on cortical temperatures and their duration: an in vitro study. Med Eng Phys. 2000 Dec;22(10):685-91. doi: 10.1016/s1350-4533(01)00016-9. PMID 11334754
- [Background] Bonfield W, Li CH. The temperature dependence of the deformation of bone. J Biomech. 1968 Dec;1(4):323-9. doi: 10.1016/0021-9290(68)90026-2. No abstract available. PMID 16329435
- [Background] Moroni A, Faldini C, Marchetti S, Manca M, Consoli V, Giannini S. Improvement of the bone-pin interface strength in osteoporotic bone with use of hydroxyapatite-coated tapered external-fixation pins. A prospective, randomized clinical study of wrist fractures. J Bone Joint Surg Am. 2001 May;83(5):717-21. doi: 10.2106/00004623-200105000-00010. PMID 11379741
- [Background] Seitz WH Jr, Froimson AI, Brooks DB, Postak P, Polando G, Greenwald AS. External fixator pin insertion techniques: biomechanical analysis and clinical relevance. J Hand Surg Am. 1991 May;16(3):560-3. doi: 10.1016/0363-5023(91)90033-8. PMID 1861045
- [Background] Ziran BH, Smith WR, Anglen JO, Tornetta P 3rd. External fixation: how to make it work. J Bone Joint Surg Am. 2007 Jul;89(7):1620-32. doi: 10.2106/JBJS.G.00425. No abstract available. PMID 17606806